CLINICAL TRIAL: NCT04918992
Title: Post-radiotherapy MRI Based AI System to Predict Radiation Proctitis for Pelvic Cancers
Brief Title: Post Radiotherapy MRI Based AI System to Predict Radiation Proctitis for Pelvic Cancers
Acronym: MRI-RP-2021
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: MRI-RP
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Pelvic Cancer
Keywords: radiation proctitis; pelvic cancers; Artificial Intelligence
MeSH Terms: conditions — Pelvic Neoplasms | interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence — investigators utilize a Artificial Intelligence (AI) supportive system to predict radiation proctitis for patients with pelvic cancers underwent radiotherapy

SUMMARY:
In this study, investigators utilize a Artificial Intelligence (AI) supportive system to predict radiation proctitis for patients with pelvic cancers underwent radiotherapy. By the system, whether the participants achieve the radiation proctitis will be identified based on the radiomics features extracted from the post radiotherapy Magnetic Resonance Imaging (MRI) . The predictive power to discriminate the radiation proctitis individuals from non-radiation proctitis patients, will be validated in this multicenter, prospective clinical study.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational clinical study for seeking out a better way to predict the radiation proctitis in patients with pelvic cancers based on the post-radiotherapy Magnetic Resonance Imaging (MRI) data. Patients who have been pathologically diagnosed as pelvic cancers will be enrolled from the Sixth Affiliated Hospital of Sun Yat-sen University, Sir Run Run Shaw Hospital and the Third Affiliated Hospital of Kunming Medical College. Patients with pelvic cancers who received radiotherapy will be enrolled and their post-radiotherapy MRI images will be used to predict their radiation proctitis or not. The clinical symptoms, endoscopic findings, imaging and histopathology as a standard. The predictive efficacy will be tested in this multicenter, prospective clinical study.

ELIGIBILITY:
Inclusion Criteria:

* pathologically diagnosed as pelvic tumours
* intending to receive or undergoing radiotherapy
* MRI (high-solution T2-weighted imaging, contrast-enhanced T1-weighted imaging, and diffusion-weighted imaging are required) examination is completed after radiotherapy

Exclusion Criteria:

* insufficient imaging quality of MRI (e.g., lack of sequence, motion artifacts)
* incomplete radiotherapy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: pelvic cancers who underwent radiotherapy will be enrolled in our study.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-06-22 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
The area under curve (AUC) of Receiver Operating Characteristic (ROC) curves of AI prediction system in prediction radiation proctitis | baseline
  The area under curve (AUC) of Receiver Operating Characteristic (ROC) curves of AI prediction system in identifying the radiation proctitis candidates from non-radiation proctitis individuals among pelvic cancers underwent radiotherapy

SECONDARY OUTCOMES:
The specificity of AI prediction system in prediction radiation proctitis | baseline
  The specificity of AI prediction system in identifying the radiation proctitis candidates from non-radiation proctitis individuals among pelvic cancers underwent radiotherapy

OTHER OUTCOMES:
The sensitivity of AI prediction system in prediction the radiation proctitis candidates | baseline
  The sensitivity of AI prediction system in identifying the radiation proctitis candidates from non-radiation proctitis individuals among pelvic cancers underwent radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Xinjuan Fan, MD, Study Chair — Sixth Affiliated Hospital, Sun Yat-sen University; Weidong Han, MD, Principal Investigator — Sir Run Run Shaw Hospital; Zhenhui Li, MD, Principal Investigator — The Third Affiliated Hospital of Kunming Medical College.
Locations (3):
- China (3):
  - the Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Kunming Medical College, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided